CLINICAL TRIAL: NCT02361684
Title: European Comparative Effectiveness Research on Internet-based Depression Treatment - Spanish Trial
Brief Title: e-Compared-S: Comparative Effectiveness Research on Internet-based Depression Treatment - Spanish Trial
Acronym: E-COMPARED_S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UJaumeI07
Record Dates: First submitted 2015-01-08; First posted 2015-02-12 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Major Depressive Disorder
Keywords: cost-effectiveness; blended treatment; Internet based treatment; Efficacy; Depression; cognitive behavioural therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blended CBT treatment (Experimental)
  Interventions: Behavioral: Blended CBT treatment
- Treatment as usual (Active Comparator)
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Blended CBT treatment — Internet based blended CBT depression treatment combines individual face-to-face cognitive behavioural therapy (CBT) with CBT delivered through an Internet based treatment platform with mobile phone components (either integrated in the treatment platform or as a separate system). The core components of the CBT treatment are: (1) psycho-education, (2) cognitive restructuring, (3) behavioural activation, (4) positive psychology, and (5) relapse prevention. These will be delivered over 10 sessions. For this study, the ratio between the number of face-to-face sessions and the number of online module will be 1/3 face-to-face and 2/3 online.
  Arms: Blended CBT treatment
Other: Treatment as usual — Treatment as usual (TAU) is defined as the routine care that subjects receive when they are diagnosed with depression in the primary care system. In practice, this means that treatment as usual may vary between patients. We will not interfere with treatment as usual but we will monitor carefully which health care services are utilized by usual care patients using patient records and through self-report
  Arms: Treatment as usual

SUMMARY:
To compare the clinical and cost-effectiveness of blended Cognitive Behavioural Therapy (CBT) for adults with major depressive disorder (MDD) with treatment as usual (TAU) in Spanish population.

DETAILED DESCRIPTION:
Depression is a common mental disorder with a negative impact on mental well-being, quality of life, and social and work-related functioning both in the short and longer term. Additionally, depression is associated with increased morbidity, mortality, health care utilization and health care costs. On a population level, depression is one of the most costly diseases. The economic costs of depression were estimated at €136.3 billion (EU25) in 2010 in the EU and are still rising. European health care systems face the challenge of improving access to cost-effective treatments while simultaneously working to sustain budgetary stability in times of economic austerity.

Internet-based depression treatment appears a very promising alternative to current routine depression treatment strategies. Meta-analyses have demonstrated the clinical effectiveness and potential cost-effectiveness of Internet-based treatment for depression in controlled research setting. Internet-based treatment thus has the potential to keep depression treatment affordable, as it enables mental health care providers to reach out to large populations needing depression treatment at a better cost-effectiveness than those of standard treatment as usual (TAU), but with similar levels of clinical efficacy and quality of care.

The trials will be conducted in 8 European countries. In Spain the trial will be carried out in routine primary, comparing the clinical and cost-effectiveness of CBT and TAU for adults with major depressive disorder (MDD). Respondents will be followed until 12 months after baseline (measures will be taken at BL, 3 months, 6 months and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Meet DSM-IV diagnostic criteria for MDD confirmed by MINI International Neuropsychiatric Interview version 5.0
* a score a score of 5 or higher on the PHQ-9 screening questionnaire.

Exclusion Criteria:

* Current high risk for suicide according to the MINI Interview section C
* Serious psychiatric co-morbidity: substance dependence, bipolar affective disorder, psychotic illness, obsessive compulsive disorder, as established at the MINI interview
* Currently receiving psychological treatment for depression in primary or specialised mental health care
* Being unable to comprehend the spoken and written language (Spanish)
* Not having access to a PC and fast Internet connection (i.e. broadband or comparable).
* Not having a Smartphone that is compatible with the mobile component of the intervention that is offered or not willing to carry a Smartphone during the duration of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 | Baseline, 3 months, 6 months and 12 months
  The PHQ-9 is a nine-item mood module that can be used to screen and to diagnose patients with depressive disorders. The 9 items are each scored on a 0-3 scale with the total score ranging from 0-27 and higher scores indicating more severe depression. The PHQ-9 has shown to have good psychometric properties (Wittkampf, Naeije, Schene, Huyser, & van Weert, 2007).

SECONDARY OUTCOMES:
Change in Quick Inventory of Depressive Symptomatology Self-Report (QIDS-16-SR) US Translation | Baseline, 3 months, 6 months and 12 months
  The QIDS is a questionnaire that screens for depressive symptoms and assesses depression severity. The QIDS is available in both clinician-rated (IDS-C) and patient self-report (IDS-SR) forms. The QIDS consists of 16 items (each item scores 0-3) and includes symptom domains of MDD based on DSM-IV and Research Diagnostic Criteria (RDC). The QIDS has shown good psychometric properties.
Change in the MINI International Neuropsychiatric Interview (M.I.N.I) version 5.0 | Baseline and 12 months
  The M.I.N.I. is a structured diagnostic interview based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and on International Classification of Diseases (ICD-10) criteria. The M.I.N.I has been translated to 65 languages and is used for both clinical and research practice. The interview compares well with Structural Clinical Interview for DSM-IV disorders (SCID) (Sheehan et al., 1998) and the Composite International Diagnostic Interview (CIDI) (Lecrubier et al., 1997; Sheehan et al., 1998).
Change in the EQ-5D-5L (EuroQol) | Baseline, 3 months, 6 months and 12 months
  The EQ-5D-5L is a self-report questionnaire which measures health related quality of life and enables conversion to utility scores to calculate Quality-Adjusted Life-Years (QALYs). The EQ-5D-5L consists of five dimensions: mobility, self-care, ordinary activities, discomfort, and mood state related to anxiety or depression. Each item consists of five categories ranging from no problems to a lot of problems (Van Agt, Essink-Bot, Krabbe, & Bonsel, 1994).
Change in the Questionnaires on Costs Associated with Psychiatric Illness (TiC-P; Hakkaart-van Rooijen, van Straten, Donker, Tiemens, 2002) | Baseline, 3 months, 6 months and 12 months
  The TiC-P is a self-report questionnaire and consists of two different parts that can be administrated separately. Part I will be used to assess the participants' healthcare utilization and medication use. Part II (short form health and labor questionnaire [SF-HLQ]) measures lost productivity costs resulting from absenteeism (being absent from work because of illness) and presenteeism (being present at work while ill which may lead to reduced efficiency) and consists of 11 items. Healthcare utilization and productivity losses will be valued using country-specific prices.
Change in the Working Alliance Inventory (WAI-SF) | 3 months
  The WAI-SF is a 12-item self-report questionnaire with responses on a 5-point Likert scale ranging from 1 (never) to 5 (always) (Hatcher & Gillaspy, 2006). The questionnaire covers three dimensions of working alliance: (1) therapeutic goals, (2) tasks, and (3) bond and the subscales have shown to have good internal consistencies. Both the patient and the 10-item therapist version of the questionnaire will be administered
Change in the credibility and expectancy questionnaire (CEQ; Devilly and Borkovec, 2000) | Baseline
  The scale consists of 6 questions, with answer options rated on a 10 point scale and on a 1-100% scale and evaluates 2 factors : credibility and expectancy
Change in the Satisfaction Questionnaire (CSQ-8; Nguyen, Attkinson, & Stegner, 1983) | 3 months
  This questionnaire is used to measure global patient satisfaction. The questionnaire consists of 8 items that are measured on a 4 points scale with total scores ranging from 8 to 32 and has shown good psychometric properties.
Change in the system usability scale (SUS; Brooke, 1996) | 3 months
  SUS is a simple ten item scale giving a global view of subjective assessments of usability of a technology system. All items are measured on a 5-point scale ranging from strongly disagree until strongly agree. Total SUS scores have a range from 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Botella Arbona, PhD, Principal Investigator — Universitat Jaume I;CIBERObn ISC III, Castellón de la Plana, Spain; Rosa Baños Rivera, PhD, Principal Investigator — Universitat de Valencia; CIBERObn ISC III, Castellón de la Plana, Spain; Azucena García-Palacios, PhD, Principal Investigator — Universitat Jaume I;CIBERObn ISC III, Castellón de la Plana, Spain; Ernestina Etchemendy, PhD, Principal Investigator — CIBERObn ISC III, Castellón de la Plana, Spain; Rocio Herrero Camarano, PhD, Principal Investigator — Universitat Jaume I
Locations (2):
- Spain (2):
  - University Jaume I, Castellon, Castellón
  - University of Valencia, Valencia

REFERENCES:
- [Background] Corruble E, Legrand JM, Zvenigorowski H, Duret C, Guelfi JD. Concordance between self-report and clinician's assessment of depression. J Psychiatr Res. 1999 Sep-Oct;33(5):457-65. doi: 10.1016/s0022-3956(99)00011-4. PMID 10504014
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] van Agt HM, Essink-Bot ML, Krabbe PF, Bonsel GJ. Test-retest reliability of health state valuations collected with the EuroQol questionnaire. Soc Sci Med. 1994 Dec;39(11):1537-44. doi: 10.1016/0277-9536(94)90005-1. PMID 7817218
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Rush AJ, Carmody T, Reimitz PE. (2000). The Inventory of Depressive Symptomatology (IDS): Clinician (IDS-C) and Self-Report (IDS-SR) ratings of depressive symptoms. International Journal of Methods in Psychiatric Research, 9(2), 45-59.
- [Background] Richardson JR, Peacock SJ, Hawthorne G, Iezzi A, Elsworth G, Day NA. Construction of the descriptive system for the Assessment of Quality of Life AQoL-6D utility instrument. Health Qual Life Outcomes. 2012 Apr 17;10:38. doi: 10.1186/1477-7525-10-38. PMID 22507254
- [Background] Pinninti NR, Madison H, Musser E, Rissmiller D. MINI International Neuropsychiatric Schedule: clinical utility and patient acceptance. Eur Psychiatry. 2003 Nov;18(7):361-4. doi: 10.1016/j.eurpsy.2003.03.004. PMID 14643565
- [Background] Nguyen TD, Attkisson CC, Stegner BL. Assessment of patient satisfaction: development and refinement of a service evaluation questionnaire. Eval Program Plann. 1983;6(3-4):299-313. doi: 10.1016/0149-7189(83)90010-1. PMID 10267258
- [Background] Lecrubier Y, Sheehan DV, Weiller E, Amorim P, Bonora I, Harnett Sheehan K, Dunbar GC. (1997). The Mini International Neuropsychiatric Interview (MINI). A short diagnostic structured interview: reliability and validity according to the CIDI. European Psychiatry, 12(5), 224-231.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Konig HH, Born A, Gunther O, Matschinger H, Heinrich S, Riedel-Heller SG, Angermeyer MC, Roick C. Validity and responsiveness of the EQ-5D in assessing and valuing health status in patients with anxiety disorders. Health Qual Life Outcomes. 2010 May 5;8:47. doi: 10.1186/1477-7525-8-47. PMID 20444251
- [Background] Hawthorne G, Richardson J, Osborne R. The Assessment of Quality of Life (AQoL) instrument: a psychometric measure of health-related quality of life. Qual Life Res. 1999 May;8(3):209-24. doi: 10.1023/a:1008815005736. PMID 10472152
- [Background] Hatcher RL, Gillaspy JA. (2007). Development and validation of a revised short version of the working alliance inventory. Psychother Res, 16:12-25.
- [Background] Hakkaart-van Rooijen L, van Straten A, Donker M, Tiemans B. (2002). Manual Trimbos/iMTA questionnaire for costs associated with psychiatric illness (TIC-P). Rotterdam: Institute for Medical Technology Assessment.
- [Background] Food Drug Administration (FDA) (1997). International conference on harmonization, good clinical practice: consolidated guidelines. Federal Register 62: 25692-25709.
- [Background] Fenwick E, O'Brien BJ, Briggs A. Cost-effectiveness acceptability curves--facts, fallacies and frequently asked questions. Health Econ. 2004 May;13(5):405-15. doi: 10.1002/hec.903. PMID 15127421
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Cuijpers P, Turner EH, Koole SL, van Dijke A, Smit F. What is the threshold for a clinically relevant effect? The case of major depressive disorders. Depress Anxiety. 2014 May;31(5):374-8. doi: 10.1002/da.22249. Epub 2014 Feb 22. PMID 24677535
- [Background] Brooke J. (1996). SUS-a quick and dirty usability scale. In Usability Eval Ind. Volume 189. Edited by Jordan PW, Thomas B, Weerdmeester BA, McClelland IL. London: Taylor & Francis Ltd; 1996:189-194.
- [Background] Black WC. The CE plane: a graphic representation of cost-effectiveness. Med Decis Making. 1990 Jul-Sep;10(3):212-4. doi: 10.1177/0272989X9001000308. PMID 2115096
- [Background] Bangor A, Kortum PT, Miller JT. (2008). An Empirical Evaluation of the System Usability Scale. Int J Hum Comput Interact 2008, 24:574-594.
- [Derived] Doukani A, Quartagno M, Sera F, Free C, Kakuma R, Riper H, Kleiboer A, Cerga-Pashoja A, van Schaik A, Botella C, Berger T, Chevreul K, Matynia M, Krieger T, Hazo JB, Draisma S, Titzler I, Topooco N, Mathiasen K, Vernmark K, Urech A, Maj A, Andersson G, Berking M, Banos RM, Araya R. Comparison of the Working Alliance in Blended Cognitive Behavioral Therapy and Treatment as Usual for Depression in Europe: Secondary Data Analysis of the E-COMPARED Randomized Controlled Trial. J Med Internet Res. 2024 May 31;26:e47515. doi: 10.2196/47515. PMID 38819882
- [Derived] van Genugten CR, Schuurmans J, Hoogendoorn AW, Araya R, Andersson G, Banos R, Botella C, Cerga Pashoja A, Cieslak R, Ebert DD, Garcia-Palacios A, Hazo JB, Herrero R, Holtzmann J, Kemmeren L, Kleiboer A, Krieger T, Smoktunowicz E, Titzler I, Topooco N, Urech A, Smit JH, Riper H. Examining the Theoretical Framework of Behavioral Activation for Major Depressive Disorder: Smartphone-Based Ecological Momentary Assessment Study. JMIR Ment Health. 2021 Dec 6;8(12):e32007. doi: 10.2196/32007. PMID 34874888
- [Derived] Vara MD, Herrero R, Etchemendy E, Espinoza M, Banos RM, Garcia-Palacios A, Lera G, Folch B, Palop-Larrea V, Vazquez P, Franco-Martin M, Kleiboer A, Riper H, Botella C. Efficacy and cost-effectiveness of a blended cognitive behavioral therapy for depression in Spanish primary health care: study protocol for a randomised non-inferiority trial. BMC Psychiatry. 2018 Mar 23;18(1):74. doi: 10.1186/s12888-018-1638-6. PMID 29566656
- [Derived] Kleiboer A, Smit J, Bosmans J, Ruwaard J, Andersson G, Topooco N, Berger T, Krieger T, Botella C, Banos R, Chevreul K, Araya R, Cerga-Pashoja A, Cieslak R, Rogala A, Vis C, Draisma S, van Schaik A, Kemmeren L, Ebert D, Berking M, Funk B, Cuijpers P, Riper H. European COMPARative Effectiveness research on blended Depression treatment versus treatment-as-usual (E-COMPARED): study protocol for a randomized controlled, non-inferiority trial in eight European countries. Trials. 2016 Aug 3;17(1):387. doi: 10.1186/s13063-016-1511-1. PMID 27488181